CLINICAL TRIAL: NCT04206280
Title: Does the Use of a Post-Operative Pedometer Affect Rate of Return of Bowel Function and Narcotic Use Following Laparoscopic Robot Assisted Radical Prostatectomy
Brief Title: Use of Pedometer Following Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB19-096
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer; Ambulation Difficulty
Keywords: radical prostatectomy; pedometer; return of bowel function; post-operative narcotic use
MeSH Terms: conditions — Prostatic Neoplasms; Mobility Limitation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pedometer group (Experimental): This group will be given a pedometer following radical prostatectomy. Subjects in the experimental group will have a graduated step-count goal as follows: POD 0-2: 2,000/day. POD 3-6: 3,000/day. POD 7-9: 4,000/day. POD 10-14: 5,000/day.
  Interventions: Behavioral: Use of a pedometer following surgery
- Control group (Active Comparator): This is the control group. Following radical prostatectomy, subjects in the control group will receive standard of care, which includes counseling regarding the importance of ambulation following surgery.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Use of a pedometer following surgery — Subjects in the study group will receive a pedometer with graduated step count goals as discussed in arm description.
  Arms: Pedometer group
Behavioral: Standard of care — Subjects in the control group will be counseled on the importance of ambulation during their pre-operative visit.
  Arms: Control group

SUMMARY:
This is a study to evaluate whether use of a pedometer following radical prostatectomy decreases post-operative narcotic use and time to return of bowel function.

DETAILED DESCRIPTION:
This is a randomized controlled prospective study looking at the effect of using a pedometer with graduated step-count goals following radical prostatectomy on return of bowel function and post-operative narcotic use. Subjects will be randomized into a control group or study group. The control group will receive standard of care, with information provided regarding the importance of ambulation following surgery. The study group will receive a pedometer with graduated step-count goals from post-operative day 0 to post-operative day 14. Both groups will be given a standardized post-operative narcotic regimen, and will be asked to record initial passage of flatus and first bowel movement. Subjects will remain on the study until initial post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

This study will include men 18-75 undergoing robot-assisted laparoscopic radical prostatectomy for prostate cancer at Virginia Mason Medical Center.

Exclusion Criteria:

* Long-term opioid use, defined by CDC as use of opioids on most days for >3 months
* History of inflammatory bowel disease
* Prior abdominopelvic radiation
* Travel to Europe during study period
* Concurrent surgery during radical prostatectomy
* Inability to ambulate
* Gastroparesis or other baseline bowel dysmotility issues
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Post operative narcotic use | 7-14 days
  Morphine equivalents used following radical prostatectomy.

SECONDARY OUTCOMES:
Rate of return of bowel function | 7-14 days
  First passage of flatus and first bowel movement following surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Corman, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No